CLINICAL TRIAL: NCT02211872
Title: An Open Phase I Single Dose Escalation Study of BI 2536 BS Administered Intravenously in Patients With Advanced Solid Tumours With Repeated Administration in Patients With Clinical Benefit
Brief Title: BI 2536 BS in Patients With Advanced Solid Tumours and Repeated Administration in Patients With Clinical Benefit
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1216.1
Record Dates: First submitted 2014-08-07; First posted 2014-08-08 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

ARMS (2):
- Treatment A (Experimental): BI 2536 BS single rising dose
  Interventions: Drug: BI 2536 BS, intravenous
- Treatment B (Experimental): BI 2536 BS multiple rising doses on three consecutive days (d1-3 schedule)
  Interventions: Drug: BI 2536 BS, intravenous

INTERVENTIONS:
Drug: BI 2536 BS, intravenous

SUMMARY:
The primary objective of this study was to determine the maximum tolerated dose (MTD) of BI 2536 BS in patients with advanced solid tumours. Secondary objectives were the evaluation of safety, efficacy, and pharmacokinetics of BI 2536 BS

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed diagnosis of advanced, non resectable and / or metastatic solid tumours, who had failed conventional treatment, or for whom no therapy of proven efficacy exists, or who were not amenable to established forms of treatment
* Evaluable tumour deposits
* Age of 18 years or older
* Life expectancy of at least 6 months
* Written informed consent consistent with international conference of harmonization (ICH) - good clinical practice (GCP) and local legislation
* Eastern Cooperative Oncology Group (ECOG, R01-0787) performance score ≤ 2
* And full recovery from all therapy-related toxicities from previous chemo-, hormone-, immuno-, or radiotherapies

Exclusion Criteria:

* Serious illness or concomitant non-oncological disease considered by the investigator to be incompatible with the trial protocol
* Pregnancy or breastfeeding
* Active infectious disease
* Known brain metastases
* Second malignancy requiring therapy
* Absolute neutrophil count less than 1500/mm3
* Platelet count less than 100 000/mm3
* Bilirubin greater than 1.5 mg/dL (> 26 μmol/L, international system of units (SI) equivalent)
* Aspartate amino transferase (AST) and / or alanine amino transferase (ALT) greater than 2.5 times the upper limit of normal (if related to liver metastases greater than five times the upper limit of normal)
* Serum creatinine greater than 1.5 mg/dL (> 132 μmol/L, SI unit equivalent)
* Sexually active women and men who are unwilling to use a medically acceptable method of contraception
* Treatment with other investigational drugs or participation in another clinical trial within the past four weeks before start of therapy or concomitantly with this trial (except for present trial drug)
* Chemo-, radio or immunotherapy within the past four weeks before start of therapy or concomitantly with this trial
* Patients unable to comply with the trial protocol
* Or active alcohol or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2004-08; Primary Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) for a single dose of BI 2536 BS | Up to 16 weeks
MTD for single doses of BI 2536 BS on 3 consecutive days | Up to 16 weeks

SECONDARY OUTCOMES:
Assessment of objective treatment response by tumour measurements | Up to 1 year
  Evaluated according to the response evaluation criteria in solid tumors (RECIST)
Number of patients with adverse events | Up to 1 year
Maximum concentration of BI 2536 BS analyte in plasma (Cmax) | Pre-dose, up to 216 hours after drug administration
Time from dosing to maximum concentration of BI 2536 BS in plasma (tmax) | Pre-dose, up to 216 hours after drug administration
Area under the concentration-time curve of BI 2536 BS in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | Pre-dose, up to 216 hours after drug administration
Percentage of the AUC0-∞ that is obtained by extrapolation (%AUC0-tz) | Pre-dose, up to 216 hours after drug administration
Terminal rate constant in plasma (λz) | Pre-dose, up to 216 hours after drug administration
Terminal half-life of BI 2536 BS in plasma (t1/2) | Pre-dose, up to 216 hours after drug administration
Mean residence time of BI 2536 BS in the body after intravenous administration (MRT) | Pre-dose, up to 216 hours after drug administration
Total clearance of BI 2536 BS in the plasma after intravascular administration (CL) | Pre-dose, up to 216 hours after drug administration
Apparent volume of distribution during the terminal phase λz following an intravascular dose (Vz) | Pre-dose, up to 216 hours after drug administration
Apparent volume of distribution at steady state following intravascular administration (Vss) | Pre-dose, up to 216 hours after drug administration
Amount of BI 2536 BS that is eliminated in urine from the time point 0 to time point 24/48 (Ae0-24/48) | Pre-dose, up to 48 hours after drug administration
Fraction of analyte eliminated in urine from time point 0 to time point 24/48 (fe0-24/48) | Pre-dose, up to 48 hours after drug administration
Renal clearance of BI 2536 BS from the time point 0 to time point 24/48 (CLR,0-24/48) | Pre-dose, up to 48 hours afterdrug administration